CLINICAL TRIAL: NCT04761900
Title: Metabolic Associated Fatty Liver Disease-simplified Definition as an Optimized Risk Stratification Tool for Predicting Metabolic Outcomes in Real World
Brief Title: MAFLD-simplified Definition as an Optimized Risk Stratification Tool for Predicting Metabolic Outcomes
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MAFLDS-1.0
Record Dates: First submitted 2021-02-13; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Metabolic Associated Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- participants were followed for the incidence of T2DM in a cohort study: performed a cohort analysis for T2DM. For incident T2DM cases, calculate the follow-up time from the date of enrollment into our study to the date of T2DM diagnosis.
  Interventions: Diagnostic Test: the differences of MAFLD and MAFLD-simplified definitions were compared in predicting metabolic diseases
- participants were followed for the incidence of hypertension in a cohort study: performed a cohort analysis for hypertension. For incident hypertension cases, calculate the follow-up time from the date of enrollment into our study to the date of hypertension diagnosis.
  Interventions: Diagnostic Test: the differences of MAFLD and MAFLD-simplified definitions were compared in predicting metabolic diseases
- participants were followed for the incidence of carotid atherosclerotic plaque in a cohort study: performed a cohort analysis for carotid atherosclerotic plaque. For incident carotid atherosclerotic plaque cases, calculate the follow-up time from the date of enrollment into our study to the date of carotid atherosclerotic plaque diagnosis.
  Interventions: Diagnostic Test: the differences of MAFLD and MAFLD-simplified definitions were compared in predicting metabolic diseases

INTERVENTIONS:
Diagnostic Test: the differences of MAFLD and MAFLD-simplified definitions were compared in predicting metabolic diseases

SUMMARY:
Recently, a consensus was proposed by an international expert panel for the terminology changed from NAFLD to Metabolic associated fatty liver disease (MAFLD). The comprehensive criteria shift to a "positive" diagnosis. It helps to increase patient awareness and understanding of fatty liver (FL), for who has high-risk metabolic dysfunction. However, a more simplified and easily applicable definition is needed. It will have an impact on clinical practice, especially in developing countries.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver diseases. It affects nearly 25% of the global population. Recently, a consensus was proposed by an international expert panel for the terminology changed from NAFLD to Metabolic associated fatty liver disease (MAFLD). The comprehensive criteria shift to a "positive" diagnosis. It helps to increase patient awareness and understanding of fatty liver (FL), for who has high-risk metabolic dysfunction. However, a more simplified and easily applicable definition is needed. It will have an impact on clinical practice, especially in developing countries. It may provide a better understanding of MAFLD, and optimize strategies for prevention of extrahepatic complications in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed ad fatty liver by ultrasound

Exclusion Criteria:

* Missing data on Ultrasound, blood glucose, BMI and metabolic status.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese adults who took annual health check-ups were enrolled in this study during 2012.
Sampling Method: Non-Probability Sample
Enrollment: 3372 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of different groups in MAFLD and MAFLD-simplified definition for the outcome of T2DM, hypertension, and carotid atherosclerotic plaque. | 7 years in a cohort study
  We performed the cohort analysis for the outcome of T2DM. T2DM was defined as the presence of any of the following conditions based on the American Diabetes Association criteria: FPG ≥126 mg/dL, HbA1c ≥6.5%; or self-reported clinician-diagnosed T2DM.

SECONDARY OUTCOMES:
Comparison of different groups in MAFLD and MAFLD-simplified definition for the outcome of hypertension | 7 years in a cohort study
  We performed the cohort analysis for the outcome of hypertension. Hypertension was defined as the presence of any of the following conditions based on Revised Chinese Guidelines for Prevention and Treatment of Hypertension in 2018: a clinic systolic BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg without the use of anti-hypertensive medications, or self-reported clinician-diagnosed hypertension.
Comparison of different groups in MAFLD and MAFLD-simplified definition for the outcome of carotid atherosclerotic plaque. | 7 years in a cohort study
  We performed the cohort analysis for the outcome of carotid atherosclerotic plaque.
  Carotid atherosclerotic plaque was assessed by recording ultrasonographic images of the right carotid artery according to Mannheim Intima-Media Thickness Consensus.

CONTACTS AND LOCATIONS:
Overall Officials: Chengfu Xu, Dr, Principal Investigator — First Affiliated Hospital of Zhejiang University

IPD SHARING:
Plan to Share IPD: Undecided